CLINICAL TRIAL: NCT02490033
Title: Randomised Trial Comparing Conventional Versus Contact Force and Electrical Coupling Index in Atrial Flutter Ablation
Brief Title: The VERISMART Trial
Acronym: VERISMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CD13/11009; 14/YH/0038 (Other: Research Ethics Committee)
Record Dates: First submitted 2015-05-18; First posted 2015-07-03 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Contact force unblinded (Other)
  Interventions: Device: Ablation Catheter
- Contact force blinded (Other)
  Interventions: Device: Ablation Catheter
- ECI unblinded (Other)
  Interventions: Device: Ablation Catheter
- ECI blinded (Other)
  Interventions: Device: Ablation Catheter

INTERVENTIONS:
Device: Ablation Catheter

SUMMARY:
Catheter ablation is now routinely used in the management of heart rhythm disorders. One of the problems with the approach is that it has not been possible to determine whether the ablation catheter is in direct contact with the heart tissue or not. This is important because too much contact has safety implications and too little means that the therapy will be ineffective. Recently two different technologies have been developed to determine contact. Currently it is not know if one is superior to the other, and the objective of this trial is to determine whether there is a difference when treating a rhythm called atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Documented paroxysmal or persistent atrial flutter

Exclusion Criteria:

* Inability or unwillingness to receive oral anticoagulation
* Previous ablation procedure for AFL
* Unwillingness or inability to complete the required follow up arrangements
* Concomitant atrial fibrillation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-04-01; Primary Completion 2017-01-06 (Actual); Study Completion 2018-10-28 (Actual)

PRIMARY OUTCOMES:
Time to achieve bi-directional block | up to 60 Seconds
  Time to achieve bi-directional block (secs) . This is defined as the time from the first lesion to the time that consistent (< one minute) bidirectional block is achieved.
  Total RF energy required for the whole procedure (sec), and total energy required for ablation (power x ablation time in secs).

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

REFERENCES:
- [Result] Begg GA, O'Neill J, Sohaib A, McLean A, Pepper CB, Graham LN, Hogarth AJ, Page SP, Gillott RG, Hill N, Walshaw J, Schilling RJ, Kanagaratnam P, Tayebjee MH. Multicentre randomised trial comparing contact force with electrical coupling index in atrial flutter ablation (VERISMART trial). PLoS One. 2019 Apr 3;14(4):e0212903. doi: 10.1371/journal.pone.0212903. eCollection 2019. PMID 30943196